CLINICAL TRIAL: NCT00463918
Title: Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Multiple-Dose Pharmacokinetics, Safety and Tolerability of Varenicline in Healthy Adolescent Smokers
Brief Title: A Phase I Study to Evaluate the Pharmacokinetics of Multiple Doses of Varenicline in Healthy Adolescent Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051070
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline
  Other Names: Chantix, Champix

SUMMARY:
This study will investigate the multiple dose pharmacokinetics, safety, and tolerability of two dose strengths of varenicline in adolescents aged 12 to 16 years who regularly smoke at least three cigarettes per day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adolescents (12 - 16 years inclusive) with a total body weight greater than 30 kg who currently smoke an average of at least 3 cigarettes per day.

Exclusion Criteria:

* Male and female subjects with a positive urine drug screen and female subjects with a positive pregnancy test.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2007-05; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: Population mean estimate for apparent plasma clearance (CL/F), central volume of distribution (V2/F) and steady-state volume of distribution (Vss/F).

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Individual predicted estimates of Cmax, Tmax, and AUCτ on Day 14 (steady-state) using the final PK model and individual post-hoc estimates of the PK parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (13):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Bardstown, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, San Antonio, Texas
- Pfizer Investigational Site, Slough, Berkshire, United Kingdom

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Fediuk DJ, Sweeney K, Sahasrabudhe V, McRae T, Byon W. Population pharmacokinetics and exposure-response analyses of varenicline in adolescent smokers. CPT Pharmacometrics Syst Pharmacol. 2021 Jul;10(7):769-781. doi: 10.1002/psp4.12645. Epub 2021 Jun 17. PMID 34062053
- [Derived] Faessel H, Ravva P, Williams K. Pharmacokinetics, safety, and tolerability of varenicline in healthy adolescent smokers: a multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Clin Ther. 2009 Jan;31(1):177-89. doi: 10.1016/j.clinthera.2009.01.003. PMID 19243716
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051070&StudyName=A%20Phase%20I%20study%20to%20evaluate%20the%20Pharmacokinetics%20of%20multiple%20doses%20of%20Varenicline%20in%20Healthy%20Adolescent%20Smokers